CLINICAL TRIAL: NCT05389670
Title: Theta-burst Repetitive Transcranial Magnetic Stimulation (TBS) of the Right Inferior Frontal Gyrus for Treatment of Nicotine Dependence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Froeliger, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2074722
Record Dates: First submitted 2021-10-25; First posted 2022-05-25 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2023-11

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous Theta-burst stimulation (cTBS) (Experimental): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Continuous TBS (cTBS) which is thought to temporarily dampen brain activity in that specific area.
  Interventions: Device: Continuous Theta-burst stimulation (cTBS)
- Sham Theta-burst stimulation (Sham Comparator)
  Interventions: Device: Sham Continuous Theta-burst stimulation (cTBS)

INTERVENTIONS:
Device: Continuous Theta-burst stimulation (cTBS) — Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Continuous TBS (cTBS) which is thought to temporarily dampen brain activity in that specific area.
  Arms: Continuous Theta-burst stimulation (cTBS)
Device: Sham Continuous Theta-burst stimulation (cTBS) — Sham cTBS, inhibitory-like patterned form of TMS.
  Arms: Sham Theta-burst stimulation

SUMMARY:
The purpose of this research study is to examine the effects of theta-burst Transcranial Magnetic Stimulation on inhibitory control and smoking among adult cigarette smokers. In a double-blind, sham controlled trial, investigators will examine the effects of 12 sessions of cTBS on executive function and smoking behavior.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 yrs. of age
2. Smoke > 5 cigarettes/day for ≥ 2 yrs, and expired carbon monoxide (CO) concentration of ≥ 8 ppm
3. English Fluency
4. Functional Vision (with corrective lenses as needed)

Exclusion Criteria:

1. Use of psychotropic and antiepileptic medications in the last month
2. Presence of an untreated illness or serious medical condition
3. History of major neurological illness
4. Contraindication to TMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for >15 min., implanted electronic device, metal in the head)
5. Any use of substances that lower seizure threshold
6. Current or past psychosis
7. Electroconvulsive therapy in last 6 months
8. Unstable cardiac disease or hypertension, severe renal or liver insufficiency, or sleep apnea
9. BAC greater than 0.0.
10. Positive urine pregnancy test
11. Any other concern that in the investigator's opinion would impact participant safety, study instruction compliance, or confound the interpretation of the study results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in the number (#) of cigarettes per day. | 2 months
  The effects of 12 sessions of continuous theta burst stimulation (cTBS) to the right inferior frontal gyrus (r.IFG) on cigarettes per day (CPD). This is measured by a core daily cigarette diary and will be measured following treatment and after making a quit attempt at: days 14, 21 and 28.
Cigarette craving scores (#) as measured by the questionnaire of smoking urges brief (QSUb). | 2 months
  The effects of 12 sessions of continuous theta burst stimulation (cTBS) to the right inferior frontal gyrus (r.IFG) on cigarette craving. This will be measured at the end of every visit to the laboratory. The Questionnaire of Smoking Urges brief (QSUb) rages from 0 to 70. Lower scores equal less craving, meaning the lower the score, the better the outcome.
Percent (%) correct on an inhibitory control GoGo/NoGo task. | 2 months
  The effects of 12 sessions of continuous theta burst stimulation (cTBS) to the right inferior frontal gyrus (r.IFG) on inhibitory control (IC) task performance. This will be measured at : baseline; after completing 12 sessions of cTBS treatment, 3-7 days following making a quit attempt and at days 14, 21 and 28 following quit attempt.
Craving regulation scores (#) on a regulation of craving task. | 2 months
  The effects of 12 sessions of continuous theta burst stimulation (cTBS) to the right inferior frontal gyrus (r.IFG) on regulation of craving (ROC) task performance. This will be measured at : baseline; after completing 12 sessions of cTBS treatment, 3-7 days following making a quit attempt and at days 14, 21 and 28 following quit attempt.

SECONDARY OUTCOMES:
Symptoms scores (#) as measured by the review of symptoms (ROS) questionnaire. | 2 months
  The safety and tolerability of 12 sessions of continuous theta burst stimulation (cTBS) to the right inferior frontal gyrus (r.IFG). This will be measured at the end of each cTBS treatment visit in the laboratory and each follow up visit. The Review of Symptoms (ROS) Questionnaire ranges from 0 to 75. Lower scores equal less symptoms, meaning the lower the score, the better the outcome.